CLINICAL TRIAL: NCT02679690
Title: Assessing Knowledge of Dietary Sodium Content and Implementation of Color-Coded Cue Cards to Aid in Improving Adherence to Low Sodium Diets in Patients With Heart Failure.
Brief Title: Assessing Knowledge of Dietary Sodium Content and Implementation of Color-Coded Cue Cards and Dietary Sodium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sheryl Ondrejko, Principal Investigator, MSN, RN, DNP Candidate, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO14110506
Record Dates: First submitted 2016-02-05; First posted 2016-02-10 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Diet, Sodium-Restricted; Heart Failure C14.280.434

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard dietary sodium education (Experimental): Standard dietary sodium education provided to patients with heart failure using voice over powerpoint presentation.
  Interventions: Behavioral: Standard Dietary Sodium Education
- color-coded cue cards (Experimental): The use of a color-coded cue cards to educate patients with heart failure on dietary sodium. The education regarding the use of the color-coded cue card was provided using a voice over powerpoint presentation.
  Interventions: Behavioral: Color-Coded Cue Cards

INTERVENTIONS:
Behavioral: Standard Dietary Sodium Education — Standard dietary education for sodium restricted diets for patients with heart failure.
  Arms: Standard dietary sodium education
Behavioral: Color-Coded Cue Cards — The use of a color-coded cue card to designate ranges of acceptable sodium content of food for comparison to labels while grocery shopping.
  Arms: color-coded cue cards

SUMMARY:
Develop an evidence-based intervention aimed at patients with heart failure (HF) using color-coded cue cards to assist in the selection of foods appropriate to their sodium restricted diet. The milligram per serving sodium content of foods will be assigned color-coded green/yellow/red designation according to very low/moderate/high as identified by the United States Food and Drug Administration's definitions of sodium content.

Assess patient knowledge of foods with sodium content appropriate for consumption on a low sodium diet before implementation of the intervention by calculating average milligrams of sodium per serving via choices made through simulated grocery store shopping.

Evaluate application of patient knowledge about low-sodium food choices using a simulated grocery store shopping intervention by calculating average milligrams of sodium per serving via choices made using the color-coded card.

DETAILED DESCRIPTION:
Each new patient referred to the heart failure (HF) clinic will be asked for their permission to participate in this project. Each patient enrolled in the project will have a random number assigned to protect identity, which will be assigned to their baseline data as well as food tally score sheets before and after intervention. Baseline data collection will include patient's sex, age,marital status, comorbidities, and education level. Using guidelines from the Centers for Disease Control (CDC) and Prevention and the Food & Drug Administration (FDA), to ensure consistency, all participating patients will be given standard dietary sodium education using a voice-over PowerPoint presentation. Approximately two weeks later, the patients will be asked to "shop" for 15 food items at a simulated grocery store. This same group of patients will then be given the evidence based intervention using a second voice-over PowerPoint presentation. During this presentation, participants will be instructed on how to use color-coded cards to assist them in choosing foods based on low/moderate/high sodium content. Green indicates foods with less than 35 mg of sodium per serving, yellow indicates foods with 35-140 mg of sodium per serving, and red indicates foods with more than 140 mg of sodium per serving. Approximately two additional weeks later, the patients will again go "shopping" for fifteen items in the same simulated grocery store using the color-coded cards that allow the patient to choose foods based on low/moderate/high sodium content. The food choices made at each grocery store encounter will be analyzed by totaling the sodium content per serving of all foods divided by the number of foods purchased (fifteen) to obtain an average milligram of sodium content per serving and then analyzed per patient, comparing that patient's pre- and post-intervention sodium per serving food choices. The average milligram of sodium per serving will be compared for each patient pre- and post-color-coded card use. The average milligrams of sodium per serving of all patients together will be totaled before the use of color-coded cards and after the use of color-coded cards. This project will assess if use of a color-coded method of dietary sodium labeling helps patients stay within their sodium restricted dietary range.

A checklist with each grocery item in the store will be used to identify and tally which products each patient chooses on each shopping trip. Each checklist will also be identified only by the assigned patient number. Staff will be instructed to provide no further dietary sodium instruction to any patient. Staff will not assist the patient in choosing grocery store items on either shopping trip, and will not comment to reinforce or discourage patient food choices during shopping.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* diagnosed with heart failure

Exclusion Criteria:

* Never participated in a heart failure clinic previously
* any patient mentally or physically unable to go grocery shopping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl A Ondrejko, MSN, Principal Investigator — University of Pittsburgh
Locations (1):
- Washington Health System Greene, Waynesburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Informed Consent Form — http://www.osiris.pitt.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Heart Failure: Patients with heart failure receiving standard dietary sodium education and then color-coded cue card education and intervention.
  Standard Dietary Sodium Education: Standard dietary education for sodium restricted diets for patients with heart failure.
  Color-Coded Cue Cards: The use of a color-coded cue card to designate ranges of acceptable sodium content of food for comparison to labels while grocery shopping.
Period: Overall Study
Arm/Group | Patients With Heart Failure
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Patient Population Pre Intervention: Patients with heart failure demographics who recieved standard dietary sodium education
Arm/Group | Patient Population Pre Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Education Level [Number; unit: participants] — Does the patient have at least a high school education as determined by asking the patient
  participants | 10

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean Milligrams of Dietary Sodium in Chosen Foods Pre- and Post- Color Coded Cue Card Intervention
Description: Each participant chose 15 grocery items at baseline (before) and after color-coded cue card dietary sodium education intervention. The outcome was the difference of the paired mean of each participant from their 15 grocery items chosen pre and post intervention.
Time Frame: two weeks and one month
Population: 9 participants who completed both PowerPoint educations and both grocery store food choices.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Patients With Heart Failure
Number analyzed (Participants) | 9
milligrams | 173.78 (61.47)

2. Secondary Outcome: Mean of Milligrams of Sodium for All Grocery Items That Were Chosen by the Total of All Participants Pre, and Post Intervention
Description: All 15 grocery items were tallied for all ten participants after the first standard dietary sodium education, with the mean obtained. This was repeated with the 9 participants who chose 15 grocery items after completing the color-coded cue card education intervention.
Time Frame: two weeks and one month
Population: The mean milligrams of sodium per serving from the 15 items of groceries chosen after standardized dietary sodium education, and then again after the education regarding the use of color-coded cue cards for dietary sodium.
Measure: Mean (Standard Deviation); unit: milligrams
Groups:
- Participants Mean Sodium Post Standard Dietary Education: Ten participants with heart failure received standard dietary sodium education and then two weeks later chose 15 items from a simulated grocery store. These 15 items were tallied for the mean milligrams of sodium per serving.
- Participants Dietary Sodium Choices Post Color-coded Cue Card: The mean milligrams of dietary sodium from the 15 grocery items chosen post color-coded cue card education intervention.
Arm/Group | Participants Mean Sodium Post Standard Dietary Education | Participants Dietary Sodium Choices Post Color-coded Cue Card
Number analyzed (Participants) | 10 | 9
milligrams | 230.3000 (65.14778) | 47.1111 (5.64456)

ADVERSE EVENTS:
Arm/Group | Patients With Heart Failure
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
* Small sample size
* a single community-based cardiology practice, a self-selected sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No